CLINICAL TRIAL: NCT06192303
Title: Prospective Study on the Efficacy and Safety of Bronchoalveolar Lavage Combined With Pathogen Metagenomic Sequencing Technology in the Diagnosis of Immune Checkpoint Inhibitor Associated Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-276
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Immune Checkpoint Inhibitor Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIP cohort
  Interventions: Diagnostic Test: Bronchoalveolar lavage and pathogen metagenomic sequencing
- non CIP cohort
  Interventions: Diagnostic Test: Bronchoalveolar lavage and pathogen metagenomic sequencing

INTERVENTIONS:
Diagnostic Test: Bronchoalveolar lavage and pathogen metagenomic sequencing — After the patient is enrolled, traditional pathogen testing will be improved, and the clinical physician will make a preliminary diagnosis based on routine pathogen testing, clinical manifestations, infection indicators, and imaging. Within 24 hours of initial diagnosis, bronchoalveolar lavage and pathogen metagenomic sequencing were performed, and BALF mNGS results were fed back to clinical physicians (without interfering with clinical decision-making). Clinical treatment data of patients were collected at 72 hours, 7 days, 14 days, and 28 days after the start of treatment, and follow-up and efficacy evaluation were conducted. Finally, a review committee consisting of two senior respiratory physicians and one imaging physician conducted a systematic review of cases to make the final diagnosis of enrolled patients (as the gold standard), analyzing the accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of BALF mNGS in diagnosing CIP.

SUMMARY:
Immune checkpoint inhibitor associated pneumonia (CIP) is a common immune related adverse reaction, accounting for 35% of all deaths. However, due to the lack of typical clinical symptoms and imaging manifestations, CIP needs to be differentiated from other diseases such as pulmonary infections and lung cancer progression. Currently, there is a lack of diagnostic gold standards, which belongs to exclusive diagnosis. Empirical diagnosis and treatment in clinical practice can easily lead to the abuse of hormones and antibiotics, and even misdiagnosis and mistreatment, resulting in patient death. Therefore, early identification of CIP and pulmonary infection is the key to successful diagnosis and treatment. The CIP diagnosis and treatment guidelines recommend performing bronchoalveolar lavage as appropriate, but there is still a lack of large-scale prospective clinical studies. The beneficial pathogen metagenomic sequencing technology for the diagnosis of pulmonary infections has not been mentioned. Our research group conducted a prospective clinical study for the first time to evaluate the effectiveness and safety of bronchoalveolar lavage combined with pathogen metagenomic sequencing technology in diagnosing CIP, explore biomarkers for diagnosing CIP, in order to improve the early diagnosis rate and treatment efficiency of CIP, and reduce the abuse of antibiotics and hormones.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form;
2. Age range from 18 to 75 years old, regardless of gender;
3. Immunosuppressive host;
4. Symptoms, signs, or imaging signs of pneumonia are visible, and empirical anti infection treatment is ineffective.

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Failure to complete microscopic examination and culture of alveolar lavage fluid or sputum;
  2. The researcher believes that there are any individuals who are not suitable for inclusion.
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity in suspected CIP patients | 2023.01-2026.01
Positive predictive value (PPV), negative predictive value (NPV) in suspected CIP patients | 2023.01-2026.01

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University Nanfang Hospital, Guangzhou, Guangdong, China